CLINICAL TRIAL: NCT02014025
Title: Laparoscopic Hepatectomy Versus Open Hepatectomy for PHC With a Tumor Size of 5-10cm:a Prospective Case-control Study
Brief Title: Laparoscopic Hepatectomy Versus Open Hepatectomy for PHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shuguo Zheng, MD (Other)
Responsible Party: Sponsor-Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG004; Zhengshuguo (Registry Identifier: Zhengshuguo)
Record Dates: First submitted 2013-12-08; First posted 2013-12-17 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Primary Liver Carcinoma
Keywords: Laparoscope hepatectomy; Open hepatectomy; large PHC; safety and sensibility
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscope hepatectomy (Experimental): We let the 45 patients who are meet the inclusion criteria .Hospital in hepatobiliary surgery E district is Group B ,they will accept laparoscopic hepatectomy: tumors are totally resected through laparoscopic.
  Interventions: Procedure: Laparoscope hepatectomy
- open hepatectomy (Experimental): We let the 45 patients who are meet the inclusion criteria .Hospital in hepatobiliary surgery A and D district is Group A ,they will accept Open Hepatectomy: tumors are totally resected by conventional laparotomy.
  Interventions: Procedure: Open hepatectomy

INTERVENTIONS:
Procedure: Open hepatectomy — We let the 45 patients who are meet the inclusion criteria .Hospital in hepatobiliary surgery A and D district is Group A ,they will accept Open Hepatectomy: tumors are totally resected by conventional laparotomy.
  Arms: open hepatectomy
Procedure: Laparoscope hepatectomy — We let the 45 patients who are meet the inclusion criteria .Hospital in hepatobiliary surgery E district is Group B ,they will accept Laparoscopic Hepatectomy: tumors are totally resected through laparoscopic.
  Arms: laparoscope hepatectomy

SUMMARY:
The purpose of this study is to compare short-term and long-term efficacy of laparoscope hepatectomy and open hepatectomy, evaluate the safety and efficacy of laparoscope hepatectomy the PHC with a tumor size of 5～10㎝,and provide class B evidence based medicine for laparoscope hepatectomy for PHC with a tumor size of 5～10㎝.

DETAILED DESCRIPTION:
Background:primary hepatic carcinoma( PHC) is the world's most common and one of the most malignant tumors, the incidence of malignant tumors in the top five in the world, second only to mortality in gastric cancer, ranked No. 3. surgery and comprehensive treatment is recognized by the medical profession Surgical approach, surgical methods include open and laparoscopic liver resection .The safety and efficacy of laparoscopic resection small PHC has been recognized, but the safety and efficacy of laparoscopy PHC resection is still a dispute, that with a tumor size of 5～10㎝, the clinical evidence is a C or D grade level from the standard definition of evidence-based medicine literature which has been published , for laparoscopic liver resection versus open liver resection for these hepatocellular carcinoma prospective case-control study has not been reported.

Intervention:We will let the 90 patients who meet the inclusion criteria .Patients in hepatobiliary surgery A, D district is undergo traditional open liver resection, hepatobiliary surgery E district is undergo laparoscopic liver resection. In addition to the surgery way is different, the rest treatments are same.

Results:

1. Clinical data include:operation time, intraoperative blood loss, volume of blood transfusion, Rate of blood transfusion, complications and mortality, postoperative liver function, resection margin, long-term curative effect and survival time were collected and analysed.
2. Statistical method:groups t-test ，univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis ，Kaplan-Meier survival analysis，Log-rank curves were used.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the Laparoscope hepatectomy group are:

  1. both male and female, aged 18 to 70;
  2. PHC diagnosis is clear preoperative;
  3. No active hepatitis and decompensated cirrhosis
  4. tumor size of 5-10 cm,no intrahepatic or distant metastasis,no tumor thrombus in the portal vein, hepatic vein, vena cava, or bile duct; and no invasion of the diaphragm or surrounding tissues;
  5. no rupture or bleeding of the tumor;
  6. Child-Pugh class A or B liver function;
  7. indocyanine green retention rate at 15 min of <15%, and a remnant liver volume/standard liver volume ratio of >50% in patients with liver cirrhosis and >35% in patients without liver cirrhosis;
  8. upper abdominal surgery, radiofrequency ablation, Transhepatic Arterial Chemotherapy And Embolization treatment, radiotherapy and chemotherapy have not been implemented and no previous surgery that absolutely contraindicated Laparoscope hepatectomy.
  9. General condition of patients and cardiopulmonary function enough to tolerate surgery
  10. voluntary participation in the study, and informed consent.
* Inclusion criteria for the Open hepatectomy group are:

meet the criteria for Laparoscope hepatectomy group;

Exclusion Criteria:

* (1) age <18 years or> 70 years , pregnant or lactating women; (2) tumor size ≥10 cm, or tumor location that would interfere with intraoperative exposure and isolation of the hepatic hilum; (3) tumor encroaching on the hepatic hilum , the portal vein, primary bile duct or tumor adjacent to the major vascular structures ; (4) unable to tolerate a pneumoperitoneum or can't tolerate surgery duo to cardiopulmonary dysfunction; (5) severe upper abdominal adhesions; (6)Pathologically confirmed positive margins

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
survival rate | 3-year
  follow-up after the surgery every 3months, to understand relapse, death, statistics 1-year, 3-year overall survival rates，disease-free survival rates , recurrence and metastasis rate.

SECONDARY OUTCOMES:
intraoperative parameters | during the operation
  operation time, intraoperative blood loss, rate of blood transfusion, tumor resection margin.

OTHER OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  ascites, pleural effusion,cardiopulmonary insufficiency,mortality, postoperative liver function failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Zhou XD, Tang ZY, Ma ZC, Wu ZQ, Fan J, Qin LX, Zhang BH. Surgery for large primary liver cancer more than 10 cm in diameter. J Cancer Res Clin Oncol. 2003 Sep;129(9):543-8. doi: 10.1007/s00432-003-0446-6. Epub 2003 Jul 30. PMID 12898232
- [Background] Jingli C, Rong C, Rubai X. Influence of colorectal laparoscopic surgery on dissemination and seeding of tumor cells. Surg Endosc. 2006 Nov;20(11):1759-61. doi: 10.1007/s00464-005-0694-4. Epub 2006 Oct 5. PMID 17024537
- [Background] Fu C, Li GY, Liu FY, Lin QH, Fang XL. [Effect of carbon dioxide pneumoperitoneum-laparoscopic surgery on tumor seeding and metastases in endometrial cancer]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2008 Feb;33(2):130-7. Chinese. PMID 18326907
- [Background] Agostini A, Robin F, Jais JP, Aggerbeck M, Vilde F, Blanc B, Lecuru F. Impact of different gases and pneumoperitoneum pressures on tumor growth during laparoscopy in a rat model. Surg Endosc. 2002 Mar;16(3):529-32. doi: 10.1007/s004640090081. Epub 2001 Nov 16. PMID 11928042
- [Background] Metzelder M, Kuebler JF, Shimotakahara A, Chang DH, Vieten G, Ure B. CO2 pneumoperitoneum increases survival in mice with polymicrobial peritonitis. Eur J Pediatr Surg. 2008 Jun;18(3):171-5. doi: 10.1055/s-2008-1038365. PMID 18493892
- [Background] Yin Z, Fan X, Ye H, Yin D, Wang J. Short- and long-term outcomes after laparoscopic and open hepatectomy for hepatocellular carcinoma: a global systematic review and meta-analysis. Ann Surg Oncol. 2013 Apr;20(4):1203-15. doi: 10.1245/s10434-012-2705-8. Epub 2012 Oct 26. PMID 23099728
- [Background] Rao A, Rao G, Ahmed I. Laparoscopic vs. open liver resection for malignant liver disease. A systematic review. Surgeon. 2012 Aug;10(4):194-201. doi: 10.1016/j.surge.2011.06.007. Epub 2011 Jul 30. PMID 22818276
- [Background] Toyosaka A, Okamoto E, Mitsunobu M, Oriyama T, Nakao N, Miura K. Intrahepatic metastases in hepatocellular carcinoma: evidence for spread via the portal vein as an efferent vessel. Am J Gastroenterol. 1996 Aug;91(8):1610-5. PMID 8759671 (Retraction: PMID 9517679 Am J Gastroenterol. 1998 Mar;93(3):492)
- [Background] Poon RT, Fan ST, Lo CM, Ng IO, Liu CL, Lam CM, Wong J. Improving survival results after resection of hepatocellular carcinoma: a prospective study of 377 patients over 10 years. Ann Surg. 2001 Jul;234(1):63-70. doi: 10.1097/00000658-200107000-00010. PMID 11420484
- [Background] Zhou XD. Recurrence and metastasis of hepatocellular carcinoma: progress and prospects. Hepatobiliary Pancreat Dis Int. 2002 Feb;1(1):35-41. PMID 14607620
- [Background] Hanazaki K, Kajikawa S, Shimozawa N, Matsushita A, Machida T, Shimada K, Yazawa K, Koide N, Adachi W, Amano J. Perioperative blood transfusion and survival following curative hepatic resection for hepatocellular carcinoma. Hepatogastroenterology. 2005 Mar-Apr;52(62):524-9. PMID 15816471
- [Background] Yeh CN, Lee WC, Jeng LB, Chen MF. Hepatic resection for hepatocellular carcinoma in Taiwan. Eur J Surg Oncol. 2002 Sep;28(6):652-6. doi: 10.1053/ejso.2002.1292. PMID 12359203
- [Background] Makino Y, Yamanoi A, Kimoto T, El-Assal ON, Kohno H, Nagasue N. The influence of perioperative blood transfusion on intrahepatic recurrence after curative resection of hepatocellular carcinoma. Am J Gastroenterol. 2000 May;95(5):1294-300. doi: 10.1111/j.1572-0241.2000.02028.x. PMID 10811342
- [Background] Kwon AH, Matsui Y, Kamiyama Y. Perioperative blood transfusion in hepatocellular carcinomas: influence of immunologic profile and recurrence free survival. Cancer. 2001 Feb 15;91(4):771-8. PMID 11241245